CLINICAL TRIAL: NCT04173962
Title: Effect of Ketamine on Laboratory-induced Stress in Healthy Subjects: A Proof-of-Concept Translational Study
Brief Title: Effect of Ketamine on Laboratory-induced Stress in Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James Murrough, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GCO 17-2440
Record Dates: First submitted 2019-11-21; First posted 2019-11-22 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers
Keywords: Ketamine; Resilience; Stress; Healthy Volunteers
MeSH Terms: interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel during the duration of the study: the ketamine arm or the midazolam arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Midazolam has similar acute anesthetic effects compared to ketamine. This makes midazolam an appropriate substance to gauge whether ketamine can affect stress response thereby acting as an active control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine group (Experimental): One 0.5mg/kg intravenous dose of ketamine
  Interventions: Drug: Ketamine
- Midazolam group (Active Comparator): One 0.045mg/kg intravenous dose of midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — administered 1 week prior to a laboratory-induced stress
  Arms: Ketamine group
Drug: Midazolam — administered 1 week prior to a laboratory-induced stress
  Arms: Midazolam group

SUMMARY:
The objective of this study is to examine the effect of a single IV dose of ketamine (0.5 mg/kg) on laboratory-induced stress in healthy participants.

DETAILED DESCRIPTION:
Stress exposure is one of the greatest risk factors for psychiatric illnesses like major depressive disorder (MDD) and post-traumatic stress disorder (PTSD). Stress resilience is the ability to experience stress without developing psychopathology. Enhancing stress resilience in at-risk populations could potentially protect against the development of stress-induced psychiatric disorders. Despite this, no resilience-enhancing pharmaceuticals have been identified yet. Pre-clinical studies showed that the administration of the glutamate N-methyl-D-aspartate (NMDA) receptor antagonist ketamine one week before an acute stress prevents the developing of depressive-like behavior in animals. In this project the study team proposes a pilot study to test if this stress prophylactic effect of ketamine applies also to humans. Ketamine will be compared to an active placebo control condition, the anesthetic midazolam, in a sample of healthy volunteers. The specific aims of this project are to test the effect of ketamine administered 1-week prior a laboratory-induced stress (1) on the positive and negative affect as measured with the Profile of Mood States (POMS) - Bipolar and (2) on the hypothalamic-pituitary-adrenal axis (HPA axis), adrenaline-noradrenaline axis (ANS axis), and self-reports of anxiety. The study team expects that subjects treated with ketamine, compared to midazolam, will experience reduced symptoms of negative affect and anxiety and a blunted hormonal response to an acute stress.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-45 years;
* Does not meet for any current or past psychiatric diagnoses as defined by DSM-V criteria;
* Participants must have a level of understanding of the English language sufficient to agree to all tests and examinations required by the study and must be able to participate fully in the informed consent process.

Exclusion Criteria:

* Any current or lifetime psychiatric disorder as determined by the Structured Clinical Interview for DSM-V Axis Disorders (SCID-5);
* Concomitant use of any medication with central nervous system activity, including treatment with antidepressants (classified as SSRIs, SNRIs, Atypical Antidepressants, TCAs);
* Any unstable medical illnesses including hepatic, renal impairment, gastroenterologic (including gastro-esophageal reflux disease), respiratory (including obstructive sleep apnea, or history of difficulty with airway management during previous anesthetics), cardiovascular (including ischemic heart disease and uncontrolled hypertension), endocrinologic, neurologic (including history of severe head injury), immunologic, or hematologic disease;
* Hypertension (systolic BP >160 mm Hg or diastolic BP >90 mm Hg) at screening or immediately prior to treatment with ketamine/midazolam;
* Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG; clinically significant is defined by an abnormality that suggests a disease and/or organ toxicity that is new or has worsened from screening, or if the abnormality is of a degree that requires additional active management (e.g., further diagnostic investigation).
* Patients who have a positive urine toxicology test for illicit substances at screening and on the treatment day.
* Previous recreational use of PCP or ketamine.
* Subjects who have received ketamine in the past.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Halloran PD, Murphy GC, Webster KE. Reliability of the bipolar form of the profile of mood states using an alternative test protocol. Psychol Rep. 2004 Oct;95(2):459-63. doi: 10.2466/pr0.95.2.459-463. PMID 15587208
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Crawford JR, Henry JD. The positive and negative affect schedule (PANAS): construct validity, measurement properties and normative data in a large non-clinical sample. Br J Clin Psychol. 2004 Sep;43(Pt 3):245-65. doi: 10.1348/0144665031752934. PMID 15333231

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted between August 2019 and March 2021 at the Icahn School of Medicine at Mount Sinai Depression and Anxiety Center for Discovery and Treatment.
Period: Overall Study
Arm/Group | Ketamine Group | Midazolam Group
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Group | Midazolam Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (7.7) | 28.2 (7.9) | 28.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 7 | 5 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in The Profile of Mood States - Bipolar Version (POMS - Bi) Composed-Anxious Subscale
Description: Change from pre- to post-TSST in The Profile of Mood States - Bipolar Version (POMS - Bi) scale measures moods and feelings primarily in clinical rather than nonclinical settings. The POMS-Bi consists of 72 adjectives that form six bipolar sub-scale scores (Composed - Anxious, Clear - Confused, Confident - Unsure, Agreeable - Hostile, Energetic - Tired, Elated - Depressed). Each of the 12 adjectives within each subscale is rated on a 4-point Likert scale with anchors of 0 = "much unlike this," 1 = "slightly unlike this," 2 = "slightly like this," and 3 = "much like this." The Composed-Anxious Subscale score is the sum of positive minus the sum of negative responses plus a constant of 18. The subscale score range is from 0 to 36. Higher score indicates higher functioning. Each subscale is separate and there is no overall score.
Time Frame: baseline and 1 week after infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Midazolam Group
Number analyzed (Participants) | 12 | 12
score on a scale | -6.8 (5.8) | -11.9 (8.6)

2. Secondary Outcome: Change in Salivary Cortisol
Description: Change from pre- to post-TSST in salivary cortisol level. Salivary cortisol level to assess effect on the hypothalamic-pituitary-adrenal axis (HPA axis).
Time Frame: baseline and 1 week after infusion
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Ketamine Group | Midazolam Group
Number analyzed (Participants) | 12 | 12
ug/dL | 0.1 (0.1) | 0.0 (0.1)

3. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change from pre- to post-TSST in Cardiovascular response to stressor during assessment visit
Time Frame: baseline and 1 week after infusion
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine Group | Midazolam Group
Number analyzed (Participants) | 12 | 12
mmHg | 4.3 (11.32) | 12.9 (11.88)

4. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change from pre- to post-TSST in Cardiovascular response to stressor during assessment visit
Time Frame: baseline and 1 week after infusion
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine Group | Midazolam Group
Number analyzed (Participants) | 12 | 12
mmHg | 4.17 (7.12) | 6.58 (6.6)

5. Secondary Outcome: Change in Heart Rate
Description: Change from pre- to post-TSST in Cardiovascular response to stressor during assessment visit
Time Frame: baseline and 1 week after infusion
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Ketamine Group | Midazolam Group
Number analyzed (Participants) | 12 | 12
beats per minute (bpm) | -0.33 (6.8) | 3.83 (7.5)

6. Secondary Outcome: Change in Salivary Alpha-amylase Level
Description: Change from pre- to post-TSST in Salivary alpha-amylase level to assess effect on the adrenaline-noradrenaline axis (ANS axis).
Time Frame: baseline and 1 week after infusion
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Ketamine Group | Midazolam Group
Number analyzed (Participants) | 12 | 12
U/mL | 109.0 (144.4) | 141.7 (106.6)

7. Secondary Outcome: Change in Positive and Negative Affect Scale (PANAS)
Description: Change from pre- to post-TSST in The Positive and Negative Affect Scale (PANAS) measures both positive and negative affect and is utilized within clinical and non-clinical populations. The PANAS is a 20-item instrument, each item is scored on a 5-likert scale from 1 (very slightly or not at all) to 5 (extremely). Positive Affect Score - total score from 10-50, with higher score indicating higher levels of positive affect. Negative Affect Score - total score from 10-50, with lower scores representing lower levels of negative affect.
Time Frame: baseline and 1 week after infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Midazolam Group
Number analyzed (Participants) | 12 | 12
score on a scale
  Negative Affect Score | 2.2 (3.7) | 4.6 (4.9)
  Positive Affect Score | -2.2 (10.1) | 1.2 (6.5)

8. Secondary Outcome: Change in Visual Analog Scale: Stressed (VAS-Stressed)
Description: Change from pre- to post-TSST in The Visual Analog Scales are scored in millimeters from the left-hand side of a 100-mm line to a perpendicular mark made by the patient at a point corresponding to the apparent magnitude of the feeling state. Full range: 0 ("not at all") to 100 ("most ever"), with higher score indicating poorer health status. The VAS-Stressed prompts participants to rate their level of stress in that exact moment on the visual analog scale.
Time Frame: baseline and 1 week after infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Midazolam Group
Number analyzed (Participants) | 12 | 12
score on a scale | 12.8 (11.6) | 12.1 (22.3)

9. Secondary Outcome: Change in Beck Anxiety Inventory (BAI)
Description: Change from pre- to post-TSST in Beck Anxiety Inventory (BAI). This is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in adults. The questions used in this measure ask about common symptoms of anxiety (such as numbness and tingling, sweating not due to heat, and fear of the worst happening). It is designed for individuals who are of 17 years of age or older and takes 5 to 10 minutes to complete. Total score range of 0-63, with higher score indicating more severe anxiety symptoms.
Time Frame: baseline and 1 week after infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Group | Midazolam Group
Number analyzed (Participants) | 12 | 12
score on a scale | 0.8 (1.4) | 2.6 (4.1)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Ketamine Group | Midazolam Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine Group (N=12) | Midazolam Group (N=12)
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT04173962/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT04173962/SAP_001.pdf